CLINICAL TRIAL: NCT06717295
Title: The CCANED-CIPHER Study: Early Cancer Detection and Treatment Response Monitoring Using AI-Based Platelet and Immune Cell Transcriptomic Profiling
Acronym: CCANED-CIPHER
Status: Recruiting | Type: Observational
Sponsor: Javier Toledo (Industry)
Responsible Party: Sponsor-Investigator, Javier Toledo, Chief Medical Officer, Dysplasia Diagnostics Limited
Organization: Dysplasia Diagnostics Limited (Industry)
Other Study IDs: CCANED-CIPHER
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Brest Cancer; Lung Cancer (NSCLC); Pancreatic Cancer, Adult; Prostate Cancers; Ovarian Cancer; Colorectal Cancer; Glioblastoma (GBM); Liver Carcinoma
Keywords: cancer screening; Liquid Biopsy; AI-based Diagnostics; Early Cancer Detection; Circulating Tumor DNA (ctDNA); RNA Profiling; Biomarker; Precision Medicine; Oncology; Health Data Analysis; Platelets; treatment response; RNA; CircRNA; Splicing; Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic cancer, adult; Prostatic Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Glioblastoma; Carcinoma, Hepatocellular; Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will utilize various biological sources to profile RNA for cancer detection and treatment response. Blood samples will be collected from all participants, serving as the source for isolating platelets and immune cells for RNA analysis.
  Platelet isolates will be extracted from these blood samples. RNA from platelets will be analyzed to identify transcriptomic profiles that may serve as biomarkers for cancer detection and monitoring. Platelets can absorb RNA from tumor cells, reflecting the cancer's molecular signature.
  In Phase 2, immune cell isolates will be separated from the blood samples of cancer patients. RNA from these immune cells will be analysed to assess transcriptomic changes associated with therapeutic responses. Known driver mutations in immune cell DNA will be assessed for correlation with RNA alterations.
  This non-invasive approach will leverage liquid biopsy methods to enhance early cancer detection and personalise treatment monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer Patients (Phase 1): This arm will include 3,500 individuals with confirmed diagnoses of common cancers such as Non-Small Cell Lung Cancer (NSCLC), Glioblastoma Multiforme (GBM), Colorectal Cancer, Hepatocellular Carcinoma (HCC), Breast Cancer, Prostate Cancer, Ovarian Cancer, and Pancreatic Cancer.
  Interventions: Diagnostic Test: DiNanoQ: A multi-cancer early detection (MCED) blood test
- Healthy Individuals: This arm will consist of 1,500 age- and sex-matched cancer-free individuals serving as controls.
  Interventions: Diagnostic Test: DiNanoQ: A multi-cancer early detection (MCED) blood test
- Cancer Patients Undergoing Treatment: This cohort will include 1,000 patients diagnosed with Hepatocellular Carcinoma (HCC) or Non-Small Cell Lung Cancer (NSCLC) across stages I to IV who are about to commence standard cancer therapy.
  Interventions: Diagnostic Test: DiNanoQ: A multi-cancer early detection (MCED) blood test; Other: DiNanoTrack: Therapeutic Response Monitoring Blood Test

INTERVENTIONS:
Diagnostic Test: DiNanoQ: A multi-cancer early detection (MCED) blood test — Procedure: Participants will undergo a single blood draw at baseline.
  Sample Analysis:
  Platelet Isolation: Platelets will be extracted from the collected blood samples.
  RNA Analysis: RNA from the isolated platelets will be extracted and analyzed using AI-based transcriptomic profiling to identify biomarkers associated with cancer.
Other: DiNanoTrack: Therapeutic Response Monitoring Blood Test — Procedures:
  Blood Sample Collection: Participants will have blood samples drawn at three time points:
  Baseline: Before therapy initiation. 6 Weeks Post-Therapy Initiation: To monitor early treatment response. 6 Months Post-Therapy Initiation: To assess longer-term therapeutic outcomes.
  Sample Analysis:
  Platelet and Immune Cell Isolation:
  Platelets: Extracted from each blood sample to continue monitoring RNA profiles.
  Immune Cells: Separated from the blood samples to analyse immune response to therapy.
  RNA Analysis:
  Platelet RNA: Analysed to observe changes in transcriptomic profiles over time using AI-based tools.
  Immune Cell RNA: Examined to assess transcriptomic changes associated with therapeutic responses.
  Data Correlation:
  Therapeutic Response Assessment: RNA profiles from platelets and immune cells will be correlated with clinical outcomes to identify biomarkers predictive of treatment efficacy, progression-free survival, relapse, and drug resistance.
  Groups: Cancer Patients Undergoing Treatment

SUMMARY:
The purpose of the CCANED-CIPHER study is to develop and validate an AI-based blood test for early cancer detection and to monitor treatment effectiveness in cancer patients. This two-phase, multi-center observational study aims to identify specific transcriptomic biomarkers in platelets and immune cells that distinguish cancer patients from healthy individuals and correlate with treatment outcomes. By analysing blood samples using artificial intelligence, the study seeks to create a safe, non-invasive method to enhance cancer diagnosis and monitor treatment responses over time.

DETAILED DESCRIPTION:
The CCANED-CIPHER study aims to revolutionise cancer diagnostics and treatment monitoring by developing and evaluating an AI-based early cancer detection tool that profiles RNA biomarkers from platelets and immune cells in blood samples. This non-invasive approach leverages liquid biopsy methods to enhance early cancer detection and provide insights into therapeutic responses.

Phase 1 (Common Cancer Early Detection [CCANED]): Early Cancer Detection

Objective:

To identify specific platelet-derived RNA biomarkers that can distinguish individuals with common cancers from healthy controls using AI-driven transcriptomic analysis.

Methodology:

* Enrol 3,500 patients with confirmed diagnoses of various common cancers and 1,500 cancer-free controls matched by age and sex.
* Obtain a single blood sample from each participant at baseline.

Laboratory Analysis:

* Platelet Isolation from blood samples.
* RNA Sequencing and transcriptomic profiling to identify RNA expression patterns.

Data Analysis:

* Use machine learning algorithms to analyse RNA data and identify biomarkers indicative of cancer presence.
* Assess sensitivity and specificity of the diagnostic tool, and evaluate its ability to differentiate between cancer types.

Expected Outcomes:

* Identification of reliable RNA biomarkers for early cancer detection.
* Validation of the AI-based diagnostic tool's accuracy and feasibility in a clinical setting.

Phase 2 ( Cancer Immuno-Profiling of Hematologic and Extracellular RNA [CIPHER]): Therapeutic Response Monitoring

Objective:

To evaluate how RNA biomarkers from immune cells and platelets correlate with therapeutic responses, providing insights into treatment efficacy and potential relapse.

Methodology:

* Enrol 1,000 cancer patients diagnosed with HCC or NSCLC across stages I to IV.
* Baseline: Collect blood samples before therapy initiation.
* Follow-Up: Additional samples at 6 weeks and 6 months post-therapy initiation.

Laboratory Analysis:

* Isolation of Immune Cells and Platelets from blood samples.
* Analysis of RNA expression changes over time.

Data Analysis:

* Evaluate associations between RNA biomarkers and clinical treatment responses.
* Develop models integrating platelet and immune cell RNA profiles to predict outcomes.

Expected Outcomes:

* Identification of biomarkers that correlate with treatment responses and progression-free survival.
* Development of predictive models for relapse and drug resistance.

Significance of the Study

The CCANED-CIPHER study addresses critical needs in oncology by providing:

* A blood test that reduces the need for invasive tissue biopsies.
* Potential for identifying cancers at an earlier, more treatable stage.
* Tailored treatment strategies based on individual biomarker profiles.
* Enhanced ability to monitor treatment effectiveness and adjust therapies accordingly.
* Early detection of relapse or drug resistance, enabling prompt clinical interventions.

Expected Impact and Future Applications: The identification of specific RNA biomarkers from platelets and immune cells has the potential to transform current practices in oncology, offering a more efficient, accurate and patient-friendly approach to cancer care.

ELIGIBILITY:
Phase 1 (Common Cancer Early Detection - CCANED)

Inclusion Criteria:

* Age: Adults aged 40 years or older.
* Confirmed diagnosis of one of the following common cancers: Non-Small Cell Lung Cancer (NSCLC), Glioblastoma Multiforme (GBM), Colorectal Cancer, Hepatocellular Carcinoma (HCC), Breast Cancer, Prostate Cancer, Ovarian Cancer, Pancreatic Cancer.

Exclusion Criteria:

* Currently pregnant.
* Presence of any active infectious diseases.
* Use of anticoagulant or antiplatelet drugs within the past 2 weeks.
* Any medical or psychological conditions that may affect the participant's ability to comply with study procedures.

Phase 2 ( Cancer Immuno-Profiling of Hematologic and Extracellular RNA - CIPHER)

Inclusion Criteria:

* Adults aged 40 years or older.
* Confirmed diagnosis of: Hepatocellular Carcinoma (HCC), Non-Small Cell Lung Cancer (NSCLC)
* Willingness to provide blood samples at the specified intervals (baseline, 6 weeks, and 6 months post-therapy initiation).

Exclusion Criteria:

* Presence of another malignancy unless it has been in remission for at least 5 years.
* Significant uncontrolled co-morbid conditions that may interfere with study participation or outcomes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The CCANED-CIPHER study will enroll a diverse, geographically dispersed population to ensure the generalizability and robustness of its findings. The study is divided into two phases, utilizing up to 10 medical centers globally across the United Kingdom (UK), Europe, America, and Asia.
  Phase 1 (CCANED):
  Participants: 5,000 adults aged 40 years or older.
  * Cancer Patients: 3,500 individuals with confirmed diagnoses of common cancers.
  * Healthy Controls: 1,500 age-matched cancer-free individuals.
  Recruitment Strategy: Participants will be identified and enrolled through the participating medical centers, ensuring a representative sample across different geographical locations.
  Phase 2 (CIPHER):
  Participants: 1,000 adults aged 40 years or older diagnosed with HCC or NSCLC across stages I to IV.
  Recruitment Strategy: Cancer patients will be recruited from the participating cancer centers, ensuring a wide representation of disease stages and treatment backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Platelet RNA Biomarkers Distinguishing Cancer Patients from Controls | Baseline (single time point)
  Utilise AI-based transcriptomic analysis of platelet RNA to identify biomarkers that differentiate between cancer patients and cancer-free controls.
Identification of RNA Biomarkers Correlating with Therapeutic Response (Phase 2) | Baseline to 6 months post-therapy initiation
  Identify RNA biomarkers from immune cells and platelets that correlate with clinical treatment response, as measured by standard criteria (e.g., RECIST)
Association Between Immune Cell Transcriptomes and AI-Based Platelet Signals | Baseline to 6 months post-therapy initiation
  Evaluate how changes in immune cell transcriptomes are associated with signals detected by the AI-based platelet profiling tool.

SECONDARY OUTCOMES:
Sensitivity and Specificity of the AI-Based Diagnostic Tool (Phase 1) | Baseline
  Calculate the diagnostic accuracy of the AI-based tool in detecting cancer among participants.
Feasibility of Platelet Transcriptomic Profiling Implementation | Phase 1 - 2 years
  Assess the practicality of sample collection, processing, and analysis in a clinical setting.
Development of Predictive Models for Treatment Outcomes (Phase 2) | Phase 2 - Two years
  Create and validate predictive models that integrate platelet and immune cell RNA profiles to predict treatment response and progression-free survival.
Identification of Biomarkers Predictive of Relapse and Drug Resistance (Phase 2) | Baseline to 6 months post-therapy initiation
  Identify RNA biomarkers predictive of relapse and drug resistance at the 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Rotimi, PhD, Study Director — Dysplasia Diagnostics Limited; Javier Toledo, Medical Degree, Principal Investigator — Dysplasia Diagnostics Limited
Locations (4):
- Various Cancer Centres, Rosario, Argentina
- NSIA- Lagos University Teaching Hospital Cancer Centre, Lagos, Nigeria
- United Kingdom (2):
  - Babraham Research Institute, Cambridge
  - Dysplasia Diagnostics Limited, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsui NB, Ng EK, Lo YM. Stability of endogenous and added RNA in blood specimens, serum, and plasma. Clin Chem. 2002 Oct;48(10):1647-53. PMID 12324479
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Smerage JB, Barlow WE, Hortobagyi GN, Winer EP, Leyland-Jones B, Srkalovic G, Tejwani S, Schott AF, O'Rourke MA, Lew DL, Doyle GV, Gralow JR, Livingston RB, Hayes DF. Circulating tumor cells and response to chemotherapy in metastatic breast cancer: SWOG S0500. J Clin Oncol. 2014 Nov 1;32(31):3483-9. doi: 10.1200/JCO.2014.56.2561. Epub 2014 Jun 2. PMID 24888818
- [Background] Siravegna G, Mussolin B, Buscarino M, Corti G, Cassingena A, Crisafulli G, Ponzetti A, Cremolini C, Amatu A, Lauricella C, Lamba S, Hobor S, Avallone A, Valtorta E, Rospo G, Medico E, Motta V, Antoniotti C, Tatangelo F, Bellosillo B, Veronese S, Budillon A, Montagut C, Racca P, Marsoni S, Falcone A, Corcoran RB, Di Nicolantonio F, Loupakis F, Siena S, Sartore-Bianchi A, Bardelli A. Clonal evolution and resistance to EGFR blockade in the blood of colorectal cancer patients. Nat Med. 2015 Jul;21(7):795-801. doi: 10.1038/nm.3870. Epub 2015 Jun 1. PMID 26030179
- [Background] Sharma SV, Lee DY, Li B, Quinlan MP, Takahashi F, Maheswaran S, McDermott U, Azizian N, Zou L, Fischbach MA, Wong KK, Brandstetter K, Wittner B, Ramaswamy S, Classon M, Settleman J. A chromatin-mediated reversible drug-tolerant state in cancer cell subpopulations. Cell. 2010 Apr 2;141(1):69-80. doi: 10.1016/j.cell.2010.02.027. PMID 20371346
- [Background] Sequist LV, Waltman BA, Dias-Santagata D, Digumarthy S, Turke AB, Fidias P, Bergethon K, Shaw AT, Gettinger S, Cosper AK, Akhavanfard S, Heist RS, Temel J, Christensen JG, Wain JC, Lynch TJ, Vernovsky K, Mark EJ, Lanuti M, Iafrate AJ, Mino-Kenudson M, Engelman JA. Genotypic and histological evolution of lung cancers acquiring resistance to EGFR inhibitors. Sci Transl Med. 2011 Mar 23;3(75):75ra26. doi: 10.1126/scitranslmed.3002003. PMID 21430269
- [Background] Redwood N, Beggs D, Morgan WE. Dissemination of tumour cells from fine needle biopsy. Thorax. 1989 Oct;44(10):826-7. doi: 10.1136/thx.44.10.826. PMID 2595626
- [Background] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Oxnard GR, Thress KS, Alden RS, Lawrance R, Paweletz CP, Cantarini M, Yang JC, Barrett JC, Janne PA. Association Between Plasma Genotyping and Outcomes of Treatment With Osimertinib (AZD9291) in Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Oct 1;34(28):3375-82. doi: 10.1200/JCO.2016.66.7162. Epub 2016 Jun 27. PMID 27354477
- [Background] Mobadersany P, Yousefi S, Amgad M, Gutman DA, Barnholtz-Sloan JS, Velazquez Vega JE, Brat DJ, Cooper LAD. Predicting cancer outcomes from histology and genomics using convolutional networks. Proc Natl Acad Sci U S A. 2018 Mar 27;115(13):E2970-E2979. doi: 10.1073/pnas.1717139115. Epub 2018 Mar 12. PMID 29531073
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Lans H, Hoeijmakers JHJ, Vermeulen W, Marteijn JA. The DNA damage response to transcription stress. Nat Rev Mol Cell Biol. 2019 Dec;20(12):766-784. doi: 10.1038/s41580-019-0169-4. Epub 2019 Sep 26. PMID 31558824
- [Background] Kucab JE, Zou X, Morganella S, Joel M, Nanda AS, Nagy E, Gomez C, Degasperi A, Harris R, Jackson SP, Arlt VM, Phillips DH, Nik-Zainal S. A Compendium of Mutational Signatures of Environmental Agents. Cell. 2019 May 2;177(4):821-836.e16. doi: 10.1016/j.cell.2019.03.001. Epub 2019 Apr 11. PMID 30982602
- [Background] Joosse SA, Beyer B, Gasch C, Nastaly P, Kuske A, Isbarn H, Horst LJ, Hille C, Gorges TM, Cayrefourcq L, Alix-Panabieres C, Tennstedt P, Riethdorf S, Schlomm T, Pantel K. Tumor-Associated Release of Prostatic Cells into the Blood after Transrectal Ultrasound-Guided Biopsy in Patients with Histologically Confirmed Prostate Cancer. Clin Chem. 2020 Jan 1;66(1):161-168. doi: 10.1373/clinchem.2019.310912. PMID 31601564
- [Background] Jackson W 3rd, Sosnoski DM, Ohanessian SE, Chandler P, Mobley A, Meisel KD, Mastro AM. Role of Megakaryocytes in Breast Cancer Metastasis to Bone. Cancer Res. 2017 Apr 15;77(8):1942-1954. doi: 10.1158/0008-5472.CAN-16-1084. Epub 2017 Feb 15. PMID 28202531
- [Background] Hustedt N, Durocher D. The control of DNA repair by the cell cycle. Nat Cell Biol. 2016 Dec 23;19(1):1-9. doi: 10.1038/ncb3452. PMID 28008184
- [Background] Hirschhaeuser F, Menne H, Dittfeld C, West J, Mueller-Klieser W, Kunz-Schughart LA. Multicellular tumor spheroids: an underestimated tool is catching up again. J Biotechnol. 2010 Jul 1;148(1):3-15. doi: 10.1016/j.jbiotec.2010.01.012. Epub 2010 Jan 25. PMID 20097238
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Background] Gay LJ, Felding-Habermann B. Contribution of platelets to tumour metastasis. Nat Rev Cancer. 2011 Feb;11(2):123-34. doi: 10.1038/nrc3004. PMID 21258396
- [Background] Diehl F, Li M, Dressman D, He Y, Shen D, Szabo S, Diaz LA Jr, Goodman SN, David KA, Juhl H, Kinzler KW, Vogelstein B. Detection and quantification of mutations in the plasma of patients with colorectal tumors. Proc Natl Acad Sci U S A. 2005 Nov 8;102(45):16368-73. doi: 10.1073/pnas.0507904102. Epub 2005 Oct 28. PMID 16258065
- [Background] Chiou YY, Hu J, Sancar A, Selby CP. RNA polymerase II is released from the DNA template during transcription-coupled repair in mammalian cells. J Biol Chem. 2018 Feb 16;293(7):2476-2486. doi: 10.1074/jbc.RA117.000971. Epub 2017 Dec 27. PMID 29282293
- [Background] Cescon DW, Bratman SV, Chan SM, Siu LL. Circulating tumor DNA and liquid biopsy in oncology. Nat Cancer. 2020 Mar;1(3):276-290. doi: 10.1038/s43018-020-0043-5. Epub 2020 Mar 20. PMID 35122035
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Best MG, Sol N, In 't Veld SGJG, Vancura A, Muller M, Niemeijer AN, Fejes AV, Tjon Kon Fat LA, Huis In 't Veld AE, Leurs C, Le Large TY, Meijer LL, Kooi IE, Rustenburg F, Schellen P, Verschueren H, Post E, Wedekind LE, Bracht J, Esenkbrink M, Wils L, Favaro F, Schoonhoven JD, Tannous J, Meijers-Heijboer H, Kazemier G, Giovannetti E, Reijneveld JC, Idema S, Killestein J, Heger M, de Jager SC, Urbanus RT, Hoefer IE, Pasterkamp G, Mannhalter C, Gomez-Arroyo J, Bogaard HJ, Noske DP, Vandertop WP, van den Broek D, Ylstra B, Nilsson RJA, Wesseling P, Karachaliou N, Rosell R, Lee-Lewandrowski E, Lewandrowski KB, Tannous BA, de Langen AJ, Smit EF, van den Heuvel MM, Wurdinger T. Swarm Intelligence-Enhanced Detection of Non-Small-Cell Lung Cancer Using Tumor-Educated Platelets. Cancer Cell. 2017 Aug 14;32(2):238-252.e9. doi: 10.1016/j.ccell.2017.07.004. PMID 28810146
- [Background] Best MG, Sol N, Kooi I, Tannous J, Westerman BA, Rustenburg F, Schellen P, Verschueren H, Post E, Koster J, Ylstra B, Ameziane N, Dorsman J, Smit EF, Verheul HM, Noske DP, Reijneveld JC, Nilsson RJA, Tannous BA, Wesseling P, Wurdinger T. RNA-Seq of Tumor-Educated Platelets Enables Blood-Based Pan-Cancer, Multiclass, and Molecular Pathway Cancer Diagnostics. Cancer Cell. 2015 Nov 9;28(5):666-676. doi: 10.1016/j.ccell.2015.09.018. Epub 2015 Oct 29. PMID 26525104
- [Background] Arroyo JD, Chevillet JR, Kroh EM, Ruf IK, Pritchard CC, Gibson DF, Mitchell PS, Bennett CF, Pogosova-Agadjanyan EL, Stirewalt DL, Tait JF, Tewari M. Argonaute2 complexes carry a population of circulating microRNAs independent of vesicles in human plasma. Proc Natl Acad Sci U S A. 2011 Mar 22;108(12):5003-8. doi: 10.1073/pnas.1019055108. Epub 2011 Mar 7. PMID 21383194
- [Background] Aitken SJ, Anderson CJ, Connor F, Pich O, Sundaram V, Feig C, Rayner TF, Lukk M, Aitken S, Luft J, Kentepozidou E, Arnedo-Pac C, Beentjes SV, Davies SE, Drews RM, Ewing A, Kaiser VB, Khamseh A, Lopez-Arribillaga E, Redmond AM, Santoyo-Lopez J, Sentis I, Talmane L, Yates AD; Liver Cancer Evolution Consortium; Semple CA, Lopez-Bigas N, Flicek P, Odom DT, Taylor MS. Pervasive lesion segregation shapes cancer genome evolution. Nature. 2020 Jul;583(7815):265-270. doi: 10.1038/s41586-020-2435-1. Epub 2020 Jun 24. PMID 32581361
- [Background] Alix-Panabieres C, Pantel K. Clinical Applications of Circulating Tumor Cells and Circulating Tumor DNA as Liquid Biopsy. Cancer Discov. 2016 May;6(5):479-91. doi: 10.1158/2159-8290.CD-15-1483. Epub 2016 Mar 11. PMID 26969689
- See also: WHO report — https://www.who.int/news-room/fact-sheets/detail/cancer